CLINICAL TRIAL: NCT06181201
Title: Association Between the Composition of the Intestinal Microbiota Before Treatment and the Tumor Response After Induction Chemotherapy Followed or Not by Neo-adjuvant Radio-chemotherapy in Locally Advanced Rectal Cancer
Brief Title: Association Between the Composition of the Intestinal Microbiota and Tumor Response in Locally Advanced Rectal Cancer
Acronym: Neo-Flo-Rect
Status: Terminated | Type: Observational
Why Stopped: Lack of eligible patients
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); L'Institut des sciences moléculaires (iSm2 UMR CNRS 7313) (Unknown)
Responsible Party: Sponsor
Other Study IDs: NéoFloRect-2201; N° Id RCB: 2022-A00572-41 (Other: ANSM)
Record Dates: First submitted 2022-12-06; First posted 2023-12-26 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cancer of Rectum
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Person with rectal cancer: People with locally advanced rectal cancer who are to receive induction chemotherapy with FLOFIRINOX followed or not by neo-adjuvant radio-chemotherapy of the Cap50 type.
  Interventions: Procedure: Stool collection

INTERVENTIONS:
Procedure: Stool collection — Stool collection is done with the "Coll-off" device (Zymo research, reference R1101-2-5) provided to the patient before and after the induction treatment and after the reference chemo-radiotherapy treatment (Cap50, Capecitabine). Collection must be carried out by the patient at home (collection using the "Coll-off" device and then transfer to a coproculture jar provided). The fresh sample is then picked up the same day by an approved transporter mandated by the promoter and will be stored at -20°C until the start of the analyses

SUMMARY:
This is an observational, single-centre study (RIPH3) for patients with rectal cancer soon to be treated with chemotherapy (+/- neo-adjuvant radio-chemotherapy) looking at the relationship between the composition of the gut microbiota before treatment and the tumour response after chemotherapy +/- radio-chemotherapy

DETAILED DESCRIPTION:
Main objective: The main objective is to test the association between :

* the gut microbiota assessed from a stool sample before the start of neoadjuvant treatment of patients (T0) on the one hand, and
* complete histological response assessed on the surgical resection specimen in patients with histologically proven stage II and III rectal tumours treated with neo-adjuvant chemotherapy followed or not by Cap50 radiochemotherapy before surgery.

Primary endpoint: The primary endpoint will be complete histological response assessed on the surgical specimen after the neoadjuvant therapy regimen. This assessment will be performed according to the usual standards and blinded to any information on the gut microbiota and on the content of short-chain fatty acids and tryptophan derivatives.

Secondary objectives:

* To explore the profile of gut microbiota composition and short-chain fatty acid content in the two groups of patients (complete histological response or not), assessed before any treatment (T0).
* To assess the changes in the composition of the intestinal flora and the content of short chain fatty acids following treatment with induction chemotherapy (T1), then preoperative radiochemotherapy (T2) if applicable, by comparison of the preoperative sample with the initial sample (T0).
* Assess the association between these taxonomic and metabolic changes (T1-T0, T2-T0) on the one hand and the histological response on the other.
* To evaluate the association between the profile of the composition of the intestinal microbiota and the content of short-chain fatty acids, as well as calprotectin (a reliable and sensitive non-invasive marker of intestinal inflammation) assessed before any treatment (T0) on the one hand, and the occurrence of toxicity during treatment, in particular digestive toxicity.

Secondary endpoints:

* Percentage of different bacteria or families of bacteria (abundance) such as Ruminococcaceae in the intestinal flora and dosage of short-chain fatty acids;
* Rarefaction curves;
* Taxonomic indicators;
* Alpha and beta diversity indices of microbiota composition;
* Determination of calprotectin by ELISA on stool sample.
* Toxicity assessed by collecting adverse events during treatment with FOLFIRINOX and for some patients during radiochemotherapy, graded according to the NCI CTCAE v5 scale and classified according to the MEDDRA dictionary;

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage II and III adenocarcinoma of the lower and middle rectum
* Patient undergoing preoperative treatment with induction chemotherapy (Folfirinox) followed or not by radio-chemotherapy of the Cap50 type
* Male or female patient aged 18 years or older
* Normal weight, overweight or moderately obese (BMI between 18.5 and 34.9)
* Patient residing in the Lille metropolitan area
* Patient affiliated to a French social protection scheme
* Patient having given his non-opposition

Exclusion Criteria:

* History of other concurrent cancers
* Presence of an intestinal (internal or external) or external urinary diversion
* Uncooperative patient for geographical, family, social or psychological reasons
* Limited legal capacity or legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with locally advanced rectal cancer who are to receive induction chemotherapy with FLOFIRINOX followed or not by neo-adjuvant radio-chemotherapy of the Cap50 type
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Gut microbiota description at T0 | at baseline
  gut microbiota assessed from a stool sample before the start of neoadjuvant treatment of patients (T0) Measurement of gut microbiota composition at T0 by high-throughput sequencing of the 16S subunit of bacterial ribosomes
histological response according to Ryan classification | after surgery, an average of 8 months after inclusion
  complete histological response assessed on the surgical resection specimen in patients with histologically proven stage II and III rectal tumours treated with neo-adjuvant chemotherapy followed or not by Cap50 radiochemotherapy before surgery and according to Ryan classification.
  TRG (TRG0-TRG3) TRG 3: extensive residual cancer with no evident tumor regression (poor or not response

CONTACTS AND LOCATIONS:
Overall Officials: Mathias CHAMAILLARD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Mehrdad JAFARI, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No